CLINICAL TRIAL: NCT02036515
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Clinical Trial to Evaluate the Safety and Efficacy of Ertugliflozin (MK-8835/PF-04971729) in the Treatment of Subjects With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin and Sitagliptin
Brief Title: Safety and Efficacy of Ertugliflozin in the Treatment of Participants With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin and Sitagliptin (MK-8835-006; VERTIS SITA2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8835-006; 2013-003697-26 (EudraCT Number); B1521015 (Other: Pfizer Study Number)
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ertugliflozin; Metformin; Sitagliptin Phosphate; glimepiride; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ertugliflozin 5 mg (Experimental): Ertugliflozin, 5 mg, oral, once daily for 52 weeks
  Interventions: Drug: Ertugliflozin 5 mg; Drug: Metformin; Drug: Sitagliptin; Drug: Glimepiride; Biological: Insulin; Drug: Placebo for ertugliflozin 10 mg
- Ertugliflozin 15 mg (Experimental): Ertugliflozin, 15 mg, oral, once daily for 52 weeks
  Interventions: Drug: Ertugliflozin 15 mg; Drug: Metformin; Drug: Sitagliptin; Drug: Glimepiride; Biological: Insulin
- Placebo (Placebo Comparator): Matching placebo to ertuglifozin, oral, once daily for 52 weeks
  Interventions: Drug: Placebo for ertugliflozin 5 mg; Drug: Metformin; Drug: Sitagliptin; Drug: Glimepiride; Biological: Insulin; Drug: Placebo for ertugliflozin 10 mg

INTERVENTIONS:
Drug: Ertugliflozin 5 mg — Ertugliflozin, oral, 5 mg tablet once daily for 52 weeks
  Other Names: MK-8835; PF-04971729
  Arms: Ertugliflozin 5 mg
Drug: Ertugliflozin 15 mg — Ertugliflozin, oral, 5 mg and 10 mg tablet once daily for 52 weeks
  Other Names: MK-8835; PF-04971729
  Arms: Ertugliflozin 15 mg
Drug: Placebo for ertugliflozin 5 mg — Matching placebo for ertugliflozin 5 mg, oral, once daily for 52 weeks
  Arms: Placebo
Drug: Metformin — Participants are to remain on their stable doses of metformin (oral, >=1500 mg/day) while receiving blinded investigational product during the double-blind treatment period.
  Other Names: Glucophage; Glucophage XR
Drug: Sitagliptin — Participants are to remain on their stable doses of sitagliptin (oral, 100 mg once daily) while receiving blinded investigational product during the double-blind treatment period.
  Other Names: JANUVIA®
Drug: Glimepiride — Glimepiride rescue medication, oral, once daily, open-label glimepiride; dose determined per the investigator's discretion
  Other Names: AMARYL
Biological: Insulin — Insulin glargine rescue medication, injectable, as required. In the event that an investigator considers use of glimepiride to not be appropriate for a participant meeting protocol specified glycemic rescue criteria, insulin glargine can be initiated as the rescue medication, and managed by the investigator according to clinical practice guidelines of the local country.
Drug: Placebo for ertugliflozin 10 mg — Matching placebo for ertugliflozin 10 mg, oral, once daily for 52 weeks
  Arms: Ertugliflozin 5 mg; Placebo

SUMMARY:
This is a safety and efficacy study of ertugliflozin (MK-8835/PF-04971729) in the treatment of participants with type 2 diabetes mellitus who have inadequate glycemic control on metformin and sitagliptin. The primary objective of the trial is to assess the hemoglobin A1C (A1C)-lowering efficacy of the addition of ertugliflozin compared to the addition of placebo with an underlying hypothesis that addition of treatment with ertugliflozin provides greater reduction in A1C compared with the addition of placebo; the primary objective will be tested for both 5-mg and 15-mg doses of ertugliflozin.

DETAILED DESCRIPTION:
The duration of the trial will be approximately 69 weeks. This will include a 1-week Screening Period, an up to 12-week wash-off/titration /dose-stabilization period, a 2-week single-blind, placebo run-in period, a 52-week double-blind, placebo-controlled treatment period (including a 26-week Phase A and 26-week Phase B), and a post-treatment telephone contact 14 days after the last dose of blinded investigational product.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus (T2DM)
* On stable diabetes therapy of metformin with either sitagliptin or another dipeptidyl peptidase-4 (DPP-4) inhibitor or a sulfonylurea (SU) prior to study participation and is willing to wash-off/switch from another DPP-4 inhibitor/SU to sitagliptin
* Body Mass Index (BMI) greater than or equal to 18.0 kg/m^2
* Male, postmenopausal female or surgically sterile female
* If a female of reproductive potential, agrees to remain abstinent or to use (or have their partner use) 2 acceptable combinations of birth control while participating in the trial and for 14 days after the last use of study drug

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis
* History of other specific types of diabetes (e.g., genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrine disorders, drug- or chemical-induced, and post-organ transplant)
* A known hypersensitivity or intolerance to any sodium-glucose co-transporter 2 (SGLT2) or DPP-4 inhibitor
* On a weight-loss program or weight-loss medication or other medication associated with weight changes and is not weight stable
* Has undergone bariatric surgery within the past 12 months or >12 months and is not weight stable
* Has been treated with insulin (except for short-term use [<= 7 days]), injectable antihyperglycemic agents (AHAs) (e.g., pramlintide, exenatide, liraglutide), pioglitazone or rosiglitazone, other sodium-glucose co-transporter 2 (SGLT2) inhibitors, alpha glucosidase inhibitors or meglitinides, bromocriptine (Cycloset™), colesevelam (Welchol™), or any other non-protocol approved AHAs within 12 weeks of study participation
* Has active, obstructive uropathy or indwelling urinary catheter
* History of myocardial infarction, unstable angina, arterial revascularization, stroke, transient ischemic attack, or New York Heart Association (NYHA) functional class III-IV heart failure within 3 months of study participation
* A history of malignancy ≤5 years prior to study participation, except for adequately treated basal or squamous cell skin cancer or in situ cervical cancer
* Known history of Human Immunodeficiency Virus (HIV)
* Has blood dyscrasias or any disorders causing hemolysis or unstable red blood cells or any other clinically significant hematological disorder (such as aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia)
* A medical history of active liver disease (other than nonalcoholic hepatic steatosis), including chronic active hepatitis B or C, primary biliary cirrhosis, or active symptomatic gallbladder disease
* Has any clinically significant malabsorption condition
* If taking thyroid replacement therapy, has not been on a stable dose for at least 6 weeks prior to study participation
* Has been previously randomized in a study with ertugliflozin
* Has participated in other studies involving an investigational drug within 30 days prior or during study participation
* Has undergone a surgical procedure within 6 weeks prior to or planned major surgery during study participation
* Has a positive urine pregnancy test
* Is pregnant or breast-feeding, or is planning to conceive during the trial, including 14 days following the last dose of study medication
* Planning to undergo hormonal therapy in preparation to donate eggs during the trial, including 14 days following the last dose of study medication
* Excessive consumption of alcoholic beverages or binge drinking
* Has donated blood or blood products within 6 weeks of study participation or plans to donate blood or blood products at any time during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2014-03-12 (Actual); Primary Completion 2016-06-06 (Actual); Study Completion 2016-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Dagogo-Jack S, Liu J, Eldor R, Amorin G, Johnson J, Hille D, Liao Y, Huyck S, Golm G, Terra SG, Mancuso JP, Engel SS, Lauring B. Efficacy and safety of the addition of ertugliflozin in patients with type 2 diabetes mellitus inadequately controlled with metformin and sitagliptin: The VERTIS SITA2 placebo-controlled randomized study. Diabetes Obes Metab. 2018 Mar;20(3):530-540. doi: 10.1111/dom.13116. Epub 2017 Oct 23. PMID 28921862
- [Derived] Gallo S, Raji A, Calle RA, Pong A, Meyer C. The effects of ertugliflozin on beta-cell function: Pooled analysis from four phase 3 randomized controlled studies. Diabetes Obes Metab. 2020 Dec;22(12):2267-2275. doi: 10.1111/dom.14149. Epub 2020 Aug 27. PMID 32700393
- [Derived] Gallo S, Calle RA, Terra SG, Pong A, Tarasenko L, Raji A. Effects of Ertugliflozin on Liver Enzymes in Patients with Type 2 Diabetes: A Post-Hoc Pooled Analysis of Phase 3 Trials. Diabetes Ther. 2020 Aug;11(8):1849-1860. doi: 10.1007/s13300-020-00867-1. Epub 2020 Jul 9. PMID 32648108
- [Derived] Patel S, Hickman A, Frederich R, Johnson S, Huyck S, Mancuso JP, Gantz I, Terra SG. Safety of Ertugliflozin in Patients with Type 2 Diabetes Mellitus: Pooled Analysis of Seven Phase 3 Randomized Controlled Trials. Diabetes Ther. 2020 Jun;11(6):1347-1367. doi: 10.1007/s13300-020-00803-3. Epub 2020 May 5. PMID 32372382
- [Derived] Liu J, Tarasenko L, Pong A, Huyck S, Wu L, Patel S, Hickman A, Mancuso JP, Gantz I, Terra SG. Efficacy and safety of ertugliflozin across racial groups in patients with type 2 diabetes mellitus. Curr Med Res Opin. 2020 Aug;36(8):1277-1284. doi: 10.1080/03007995.2020.1760228. Epub 2020 May 13. PMID 32324082
- [Derived] Liu J, Tarasenko L, Pong A, Huyck S, Patel S, Hickman A, Mancuso JP, Ellison MC, Gantz I, Terra SG. Efficacy and safety of ertugliflozin in Hispanic/Latino patients with type 2 diabetes mellitus. Curr Med Res Opin. 2020 Jul;36(7):1097-1106. doi: 10.1080/03007995.2020.1760227. Epub 2020 May 13. PMID 32324065
- [Derived] Liu J, Patel S, Cater NB, Wu L, Huyck S, Terra SG, Hickman A, Darekar A, Pong A, Gantz I. Efficacy and safety of ertugliflozin in East/Southeast Asian patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2020 Apr;22(4):574-582. doi: 10.1111/dom.13931. Epub 2020 Jan 3. PMID 31797522
- [Derived] Liu J, Pong A, Gallo S, Darekar A, Terra SG. Effect of ertugliflozin on blood pressure in patients with type 2 diabetes mellitus: a post hoc pooled analysis of randomized controlled trials. Cardiovasc Diabetol. 2019 May 7;18(1):59. doi: 10.1186/s12933-019-0856-7. PMID 31064361

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were randomized to Ertugliflozin 15 mg, but did not receive any treatment.
Period: Overall Study
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Started | 156 | 155 | 153
Treated | 156 | 153 | 153
Completed | 151 | 143 | 139
Not Completed | 5 | 12 | 14
Not completed — Adverse Event | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Non-compliance with study drug | 0 | 0 | 2
Not completed — Screen failure | 0 | 2 | 0
Not completed — Withdrawal by Subject | 4 | 7 | 9
Not completed — Hyperglycemia | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants as treated population excludes two participants randomized to Ertugliflozin 15 mg but did not receive any treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo | Total
Number analyzed (Participants) | 156 | 153 | 153 | 462
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.2 (9.3) | 59.7 (8.6) | 58.3 (9.2) | 59.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 71 | 53 | 199
  Male | 81 | 82 | 100 | 263
Hemoglobin A1c (A1C) [Mean (Standard Deviation); unit: Percent] — Participants with baseline data: ertugliflozin 5 mg, n=155; ertugliflozin 15 mg, n=152; placebo, n=152; total, n=459
  Percent | 8.05 (0.86) | 8.00 (0.83) | 8.03 (0.93) | 8.03 (0.88)
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dL] — Participants with baseline data: ertugliflozin 5 mg, n=156; ertugliflozin 15 mg, n=152; placebo, n=152; total, n=460
  mg/dL | 167.7 (37.7) | 171.7 (39.1) | 169.6 (37.8) | 169.7 (38.2)
Body weight [Mean (Standard Deviation); unit: Kilograms] | 87.6 (18.6) | 86.6 (19.5) | 86.4 (20.8) | 86.9 (19.6)
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 87.0 (17.5) | 86.9 (15.6) | 89.9 (17.5) | 87.9 (16.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C at Week 26
Description: A1C is measured as percent. Thus this change from baseline reflects the Week 26 A1C percent minus the Week 0 A1C percent. Laboratory measurements were performed after an overnight fast ≥10 hours in duration. Data presented exclude data following the initiation of rescue therapy.
Time Frame: Baseline and Week 26
Population: Analysis population included all randomized participants who took at least one dose of study medication and had at least one A1C measurement (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 153
Percent | -0.78 [-0.91 to -0.65] | -0.86 [-0.99 to -0.72] | -0.09 [-0.23 to -0.04]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; Model is fitted with effects for treatment, time, interaction of time by treatment, effects for baseline eGFR and prior antihyperglycemic medication; Difference in least squares mean = -0.69, 95% CI 2-sided [-0.87 to -0.50]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; p < 0.001, cLDA; [statistical method as in outcome 1, analysis 1]; Difference in least squares mean = -0.76, 95% CI 2-sided [-0.95 to -0.58]

2. Primary Outcome: Percentage of Participants Experiencing An Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with this treatment. Data presented include data following the initiation of rescue therapy.
Time Frame: Up to Week 54
Population: Analysis population consisted of all randomized participants who took at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 153
Percentage of participants | 57.7 | 60.1 | 63.4
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; Difference in percentage = -5.7, 95% CI 2-sided [-16.5 to 5.2]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; Difference in percentage = -3.3, 95% CI 2-sided [-14.1 to 7.6]

3. Primary Outcome: Percentage of Participants Discontinuing Study Treatment Due to an AE
Description: as for outcome 2
Time Frame: Up to Week 52
Population: Analysis population consisted of all randomized participants who took at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 153
Percentage of participants | 4.5 | 3.9 | 3.9
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; Difference in percentage = 0.6, 95% CI 2-sided [-4.4 to 5.6]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; Difference in percentage = 0.0, 95% CI 2-sided [-4.9 to 4.9]

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26
Description: The change from baseline is the Week 26 FPG minus the Week 0 FPG. Laboratory measurements were performed after an overnight fast ≥10 hours in duration. Data presented exclude data following the initiation of rescue therapy.
Time Frame: Baseline and Week 26
Population: Analysis population included all randomized participants who took at least one dose of study medication and had at least one FPG measurement (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 153
mg/dL | -26.91 (-32.58) [-32.58 to -21.24] | -33.04 [-38.71 to -27.36] | -1.76 [-7.70 to 4.18]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, cLDA; [statistical method as in outcome 1, analysis 1]; Differenc in least squares means = -25.15, 95% CI 2-sided [-32.76 to -17.54]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; p < 0.001, cLDA; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -31.28, 95% CI 2-sided [-38.90 to -23.66]

5. Secondary Outcome: Change From Baseline in Body Weight at Week 26
Description: The change from baseline is the Week 26 body weight minus the Week 0 body weight. Data presented exclude data following the initiation of rescue therapy.
Time Frame: Baseline and Week 26
Population: Analysis population included all randomized participants who took at least one dose of study medication and had at least one body weight measurement (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 153
kg | -3.35 [-3.78 to -2.91] | -3.04 [-3.48 to -2.60] | -1.32 [-1.77 to -0.87]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, cLDA; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -2.03, 95% CI 2-sided [-2.65 to -1.40]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; p < 0.001, cLDA; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -1.72, 95% CI 2-sided [-2.35 to -1.09]

6. Secondary Outcome: Percentage of Participants With an A1C <7% (53 mmol/Mol) at Week 26
Description: A1C is measured as percent. Laboratory measurements were performed after an overnight fast ≥10 hours in duration. Data presented exclude data following the initiation of rescue therapy.
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 153
Percentage of participants | 32.1 | 39.9 | 17.0
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Logistic regression model fitted with terms for treatment, baseline A1C, baseline eGFR and prior antihyperglycemic medication; Odds Ratio (OR) = 3.16, 95% CI 2-sided [1.74 to 5.72]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 6, analysis 1]; Difference in least squares means = 4.43, 95% CI 2-sided [2.44 to 8.02]

7. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure at Week 26
Description: The change from baseline is the Week 26 systolic blood pressure minus the Week 0 systolic blood pressure. Sitting blood pressure was measured in triplicate. Data presented exclude data following the initiation of rescue therapy.
Time Frame: Baseline and Week 26
Population: Analysis population included all randomized participants who took at least one dose of study medication and had at least one systolic blood pressure measurement (baseline or post-baseline).
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 153
mmHg
  Baseline | 130.87 (0.62) [-5.52 to -2.09] | 130.87 (0.62) [-6.55 to -3.09] | 130.87 (0.62) [-2.70 to 0.94]
  Change from baseline | -3.81 (0.87) | -4.82 (0.88) | -0.88 (0.93)
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.019, cLDA; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -2.93, 95% CI 2-sided [-5.36 to -0.49]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; p = 0.002, cLDA; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -3.94, 95% CI 2-sided [-6.39 to -1.50]

8. Secondary Outcome: Change From Baseline in Hemoglobin A1C at Week 52
Description: A1C is measured as percent. Thus this change from baseline reflects the Week 52 A1C percent minus the Week 0 A1C percent. Laboratory measurements were performed after an overnight fast ≥10 hours in duration. Data presented exclude data following the initiation of rescue therapy.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 153
Percent | -0.75 [-0.90 to -0.59] | -0.81 [-0.97 to -0.66] | 0.02 [-0.15 to 0.19]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = -0.76, 95% CI 2-sided [-0.98 to -0.54]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = -0.83, 95% CI 2-sided [-1.05 to -0.61]

9. Secondary Outcome: Change From Baseline in FPG at Week 52
Description: The change from baseline is the Week 52 FPG minus the Week 0 FPG. Laboratory measurements were performed after an overnight fast ≥10 hours in duration. Data presented exclude data following the initiation of rescue therapy.
Time Frame: Baseline and Week 52
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 153
mg/dL | -25.57 [-30.91 to -20.23] | -26.38 [-31.80 to -20.97] | 3.19 [-3.08 to 9.47]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = -28.76, 95% CI 2-sided [-36.44 to -21.09]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = -29.58, 95% CI 2-sided [-37.30 to -21.85]

10. Secondary Outcome: Change From Baseline in Body Weight at Week 52
Description: The change from baseline is the Week 52 body weight minus the Week 0 body weight. Data presented exclude data following the initiation of rescue therapy.
Time Frame: Baseline and Week 52
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 153
kg | -3.46 [-4.07 to -2.85] | -2.83 [-3.45 to -2.21] | -0.95 [-1.65 to -0.26]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = -2.51, 95% CI 2-sided [-3.43 to -1.59]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = -1.88, 95% CI 2-sided [-2.81 to -0.95]

11. Secondary Outcome: Percentage of Participants With an A1C <7% (53 mmol/Mol) at Week 52
Description: as for outcome 6
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 153
Percentage of participants | 33.3 | 32.7 | 13.7
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; Odds Ratio (OR) = 3.63, 95% CI 2-sided [1.98 to 6.64]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; Odds Ratio (OR) = 4.02, 95% CI 2-sided [2.22 to 7.28]

12. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure at Week 52
Description: The change from baseline is the Week 52 systolic blood pressure minus the Week 0 systolic blood pressure. Sitting blood pressure was measured in triplicate. Data presented exclude data following the initiation of rescue therapy.
Time Frame: Baseline and Week 52
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 153
mmHg
  Baseline | 130.92 (0.62) [-6.03 to -2.29] | 130.92 (0.62) [-5.98 to -2.20] | 130.92 (0.62) [-1.41 to 3.06]
  Change from baseline | -4.16 (0.95) | -4.09 (0.96) | 0.83 (1.14)
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = -4.99, 95% CI 2-sided [-7.82 to -2.15]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = -4.92, 95% CI 2-sided [-7.76 to -2.07]

13. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure at Week 26
Description: The change from baseline is the Week 26 diastolic blood pressure minus the Week 0 diastolic blood pressure. Sitting blood pressure was measured in triplicate. Data presented exclude data following the initiation of rescue therapy.
Time Frame: Baseline and Week 26
Population: Analysis population included all randomized participants who took at least one dose of study medication and had at least one diastolic blood pressure measurement (baseline or post-baseline).
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 153
mmHg
  Baseline | 78.42 (0.36) [-2.88 to -0.48] | 78.42 (0.36) [-3.02 to -0.60] | 78.42 (0.36) [-1.71 to 0.84]
  Change from baseline | -1.68 (0.61) | -1.81 (0.62) | -0.43 (0.65)
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = -1.24, 95% CI 2-sided [-2.97 to 0.48]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = -1.38, 95% CI 2-sided [-3.11 to 0.36]

14. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure at Week 52
Description: The change from baseline is the Week 52 diastolic blood pressure minus the Week 0 diastolic blood pressure. Sitting blood pressure was measured in triplicate. Data presented exclude data following the initiation of rescue therapy.
Time Frame: Baseline and Week 52
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 153
mmHg
  Baseline | 78.44 (0.36) [-2.72 to -0.32] | 78.44 (0.36) [-2.59 to -0.17] | 78.44 (0.36) [-1.97 to 0.91]
  Change from baseline | -1.52 (0.61) | -1.38 (0.62) | -0.53 (0.73)
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = -0.99, 95% CI 2-sided [-2.82 to 0.84]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = -0.85, 95% CI 2-sided [-2.69 to 0.99]

15. Secondary Outcome: Percentage of Participants Receiving Glycemic Rescue Medication by Week 26
Description: Glycemic rescue medication was initiated for participants who met progressively more stringent glycemic rescue criteria. Rescue medication included glimepiride (or insulin glargine if glimepiride was not considered appropriate for the participant).
Time Frame: Week 26
Population: Analysis population included all randomized participants who took at least one dose of trial treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 153
Percentage of participants | 1.3 | 2.0 | 16.3
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; Difference in percent = -15.1, 95% CI 2-sided [-21.9 to -9.4]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; Difference in percent = -14.4, 95% CI 2-sided [-21.3 to -8.5]

16. Secondary Outcome: Percentage of Participants Receiving Glycemic Rescue Medication by Week 52
Description: as for outcome 15
Time Frame: Week 52
Population: Analysis population included all randomized participants who took at least one dose of trial treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 153
Percentage of participants | 12.8 | 13.7 | 41.8
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; Difference in percentage = -29.0, 95% CI 2-sided [-38.3 to -19.4]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; Difference in percentage = -28.1, 95% CI 2-sided [-37.5 to -18.4]

17. Secondary Outcome: Time to Initiation of Glycemic Rescue by Week 26
Description: Glycemic rescue medication was initiated for participants who met progressively more stringent glycemic rescue criteria. Rescue medication included glimepiride (or insulin glargine if glimepiride was not considered appropriate for the participant). Data presented are the minimum and maximum times to the initiation of rescue therapy in days. Below data include data from 1 participant in the Placebo arm who continued Phase A treatment for an additional 30 days.
Time Frame: Up to Week 26 (plus 30 days for 1 placebo participant)
Population: Analysis population included all randomized participants who took at least one dose of trial treatment
Measure: Number; unit: Days
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 153
Days
  Minimum time to initiation of glycemic rescue | 135 | 43 | 26
  Maximum time to initiation of glycemic rescue | 141 | 147 | 212

18. Secondary Outcome: Time to Initiation of Glycemic Rescue by Week 52
Description: Glycemic rescue medication was initiated for participants who met progressively more stringent glycemic rescue criteria. Rescue medication included glimepiride (or insulin glargine if glimepiride was not considered appropriate for the participant). Data presented are the minimum and maximum times to the initiation of rescue therapy in days.
Time Frame: Up to week 52
Population: Analysis population included all randomized participants who took at least one dose of trial treatment.
Measure: Number; unit: Days
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 153
Days
  Minimum time to initiation of glycemic rescue | 135 | 43 | 26
  Maximum time to initiation of glycemic rescue | 295 | 299 | 327

19. Secondary Outcome: Baseline Homeostasis Model Assessment of β-cell Function (HOMA-%β) Value
Description: HOMA-%β is a well-accepted means of assessing fasting β-cell function, and is calculated using measured C-peptide and glucose levels and is measured as a percentage of a normal reference population. HOMA-%β = [20 x fasting insulin (μU/mL)] / [fasting plasma glucose (mmol/L) - 3.5]
Time Frame: Baseline
Population: Analysis population included all randomized participants who took at least one dose of study medication and had HOMA-%β measurement at baseline.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 140 | 131 | 127
Percentage | 47.99 (23.890) [8.87 to 17.68] | 48.54 (34.782) [7.94 to 16.93] | 48.04 (30.733) [-4.08 to 5.12]

20. Secondary Outcome: Change From Baseline in HOMA-%β at Week 26
Description: HOMA-%β is a well-accepted means of assessing fasting β-cell function, and is calculated using measured C-peptide and glucose levels and is measured as a percentage of a normal reference population. HOMA-%β = [20 x fasting insulin (μU/mL)] / [fasting plasma glucose (mmol/L) - 3.5]. Data presented exclude data following the initiation of rescue therapy.
Time Frame: Baseline and Week 26
Population: Analysis population included all randomized participants who took at least one dose of study medication and had at least one HOMA-%β measurement (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 153 | 151 | 147
Percentage | 13.28 [8.87 to 17.68] | 12.43 [7.94 to 16.93] | 0.52 [-4.08 to 5.12]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = 12.75, 95% CI 2-sided [6.83 to 18.68]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = 11.91, 95% CI 2-sided [5.94 to 17.88]

21. Secondary Outcome: Change From Baseline in HOMA-%β at Week 52
Description: as for outcome 20
Time Frame: Baseline and Week 52
Population: as for outcome 20
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 155 | 152 | 152
Percentage | 10.85 [6.29 to 15.41] | 10.93 [6.24 to 15.61] | -1.93 [-6.88 to 3.02]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = 12.78, 95% CI 2-sided [6.54 to 19.03]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = 12.86, 95% CI 2-sided [6.54 to 19.18]

22. Secondary Outcome: Baseline EQ-5D 3-level Version (EQ-5D-3L) Questionnaire Score
Description: The EQ-5D-3L is a health profile questionnaire that assesses quality of life along 5 dimensions. Participants rate 5 aspects of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) by choosing from 3 answering options (1=no problems; 2=some problems; 3=extreme problems). The summed score ranges from 1-15 with "3" corresponding to no problems and "15" corresponding to severe problems in the 5 dimensions. EQ-5D-3L also includes an EQ visual analogue score (VAS) that ranges between 100 (best imaginable health) and 0 (worst imaginable health). Total index EQ-5D-3L summary score is weighted with a range of -0.594 (worst) to 1.0 (best).
Time Frame: Baseline
Population: Analysis population included all randomized participants who took at least one dose of study medication and had a baseline EQ-5D-3L measurement.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 150 | 150 | 152
Score on a scale | 0.88 (0.166) [-0.02 to 0.03] | 0.89 (0.182) [-0.00 to 0.04] | 0.90 (0.144) [-0.01 to 0.04]

23. Secondary Outcome: Change From Baseline in EQ-5D-3L Questionnaire Score at Week 26
Description: The EQ-5D-3L is a health profile questionnaire that assesses quality of life along 5 dimensions. Participants rate 5 aspects of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) by choosing from 3 answering options (1=no problems; 2=some problems; 3=extreme problems). The summed score ranges from 3-15 with "3" corresponding to no problems and "15" corresponding to severe problems in the 5 dimensions. EQ-5D-3L also includes an EQ VAS that ranges between 100 (best imaginable health) and 0 (worst imaginable health). Decrease from baseline in EQ-5D-3L signifies improvement. Total index EQ-5D-3L summary score is weighted with a range of -0.594 (worst) to 1.0 (best). Data presented exclude data following the initiation of rescue therapy.
Time Frame: Baseline and Week 26
Population: Analysis population included all randomized participants who took at least one dose of study medication and had at least one EQ-5D-3L measurement (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 155 | 151 | 153
Score on a scale | 0.00 [-0.02 to 0.03] | 0.02 [-0.00 to 0.04] | 0.01 [-0.01 to 0.04]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = -0.01, 95% CI 2-sided [-0.04 to 0.02]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = 0.01, 95% CI 2-sided [-0.02 to 0.04]

24. Secondary Outcome: Change From Baseline in EQ-5D-3L Score at Week 52
Description: as for outcome 23
Time Frame: Baseline and Week 52
Population: as for outcome 23
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 155 | 151 | 153
Score on a scale | 0.03 [-0.00 to 0.05] | -0.00 [-0.03 to 0.03] | 0.02 [-0.01 to 0.06]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = 0.00, 95% CI 2-sided [-0.04 to 0.04]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; Difference in least squares means = -0.02, 95% CI 2-sided [-0.07 to 0.02]

ADVERSE EVENTS:
Time Frame: Up to 54 weeks
Description: Data presented below includes data following the initiation of rescue therapy for the entire study (ie, all data after randomization, with no upper limit on the follow-up window for participants who discontinued study drug). Two participants randomized to ertugliflozin 15 mg didn't receive any study medication & aren't included in the below tables
Groups:
- Ertugliflozin 5 mg (Phase A+B): Ertugliflozin, 5 mg, oral, once daily for 52 weeks
- Ertugliflozin 15 mg (Phase A+B): Ertugliflozin, 15 mg, oral, once daily for 52 weeks
- Placebo (Phase A+B): Matching placebo to ertuglifozin, oral, once daily for 52 weeks
Arm/Group | Ertugliflozin 5 mg (Phase A+B) | Ertugliflozin 15 mg (Phase A+B) | Placebo (Phase A+B)
Serious Adverse Events (participants affected / at risk) | 13/156 | 3/153 | 8/153
Other Adverse Events (participants affected / at risk) | 24/156 | 18/153 | 29/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertugliflozin 5 mg (Phase A+B) (N=156) | Ertugliflozin 15 mg (Phase A+B) (N=153) | Placebo (Phase A+B) (N=153)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bone tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis tuberculous (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bening ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertugliflozin 5 mg (Phase A+B) (N=156) | Ertugliflozin 15 mg (Phase A+B) (N=153) | Placebo (Phase A+B) (N=153)
Nasopharyngitis (Infections and infestations) | 8 (8) | 6 (6) | 5 (6)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (5) | 8 (9)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (16) | 5 (11) | 11 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.